CLINICAL TRIAL: NCT01710462
Title: Clinical Study, Multicenter, Randomized With 2 Arms of Pantoprazole + Domperidone and Pantoprazole Isolated at the Gastroesophageal Reflux Disease
Acronym: PANDA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Change of company's strategy
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EF129
Record Dates: First submitted 2012-10-15; First posted 2012-10-19 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2012-10

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole; Domperidone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pantoprazole + Domperidone (Experimental): The combination of pantoprazole and domperidone provided for the study will be the new incremental formulation produced by Eurofarma. For this study will be used doses of capsules containing 20 mg pantoprazole, 20 mg of domperidone.
  Interventions: Drug: Pantoprazole + Domperidone
- Pantozol® (Takeda) (Active Comparator): The Pantozol® may be presented in boxes of coated tablets of 20 mg or 40 mg. For this study will be used 20 mg tablets.
  Interventions: Drug: Pantozol®

INTERVENTIONS:
Drug: Pantoprazole + Domperidone
  Arms: Pantoprazole + Domperidone
Drug: Pantozol®
  Arms: Pantozol® (Takeda)

SUMMARY:
This superiority phase III study to compare the combination of Pantoprazole and Domperidone with Pantoprazole isolated to the treatment of gastroesophageal reflux disease. The hypothesis is that combination of the two medication at the unique capsule is better to the patients because decrease the quantity of times the patients need to take medicines during the day.

ELIGIBILITY:
Inclusion Criteria:

1. Subscription of IC;
2. Age ≥ 18 years and <70 years
3. Diagnosis initial clinical or previous symptomatic GERD;
4. Symptom score ≥ 4;
5. Ability to conduct examinations of endoscopy;
6. Ability to perform washout of drug classes PPIs, H2 antagonists, and prokinetics for at least 14 days.

Exclusion Criteria:

1. Presence of esophagitis requiring intervention, esophageal varices, Barrett's esophagus, scleroderma, ulcers (gastric or duodenal), atrophic gastritis, or vagotomy pangastritis detected at the time of study enrollment;
2. Eradication treatment of H. pylori completed less than 15 days of V0;
3. Presence of alarm symptoms (weight loss greater than 5% in the last 60 days, no evidence of gastrointestinal bleeding);
4. Gastric or esophageal surgery prior (except for simple ulcer closure);
5. Females in pregnancy, lactation, or who wish to become pregnant if they refuse to use adequate contraception during the study period.
6. Concomitant serious diseases such as kidney failure, heart and liver;
7. Suspected or confirmed any cancer except carcinoma in situ or nonmelanoma skin cancer diagnosed in the last 5 years;
8. History of gastric cancer in relatives of 1st degree;
9. Use of illicit drugs or alcohol abuse according to the investigator;
10. Values changed (outside the normal range for the local laboratory) in leukocytes, platelets or hemoglobin;
11. Significant changes in serum sodium, potassium, calcium or creatinine;
12. Intolerance or allergy to any component of the drugs evaluated in the study;
13. Use of anti-inflammatory drugs (NSAIDs), antiemetics, macrolides and systemic steroids for a period of not less than 2 weeks prior to the study or who have expected necessity of prolonged use during the study treatment;
14. Current use of bisphosphonates, as well as those who need calcium channel blockers or other drugs that affect esophageal motility or lower esophageal sphincter tone.
15. Use of other scheduled medications metabolized by cytochrome CYP3A4 during the study;
16. Participation recent (past 12 months) or participation in a clinical trial expected during this study in other clinical trials involving drugs of any kind.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08

PRIMARY OUTCOMES:
Evaluate the efficacy of pantoprazole + domperidone Eurofarma at the treatment of gastroesophageal reflux disease in relation to the reference drug during 56 days using the score of symptoms | Evaluation at the gastroesophageal reflux disease in 56 treatment days
  The primary objective of the study is to evaluate the efficacy of combining incremental pantoprazole and domperidone Eurofarma the treatment of gastroesophageal reflux disease in relation to the reference drug. The primary endpoint is the score of symptoms (heartburn and regurgitation) including the severity and frequency after treatment

SECONDARY OUTCOMES:
Quality of life during the study treatment | Evaluation at the gastroesophageal reflux disease in 56 treatment days
Endoscopic cure rate for patients with erosive gastroesophageal reflux disease | Evaluation at the gastroesophageal reflux disease in 56 treatment days
Frequency of adverse events observed | Evaluation at the gastroesophageal reflux disease in 56 treatment days

CONTACTS AND LOCATIONS:
Locations (8):
- Brazil (8):
  - Goiania, Goiânia, Goiás
  - Belo Horizonte, Belo Horizonte, Minas Gerais
  - Curitiba, Curitiba, Paraná
  - Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Campinas, Campinas, São Paulo
  - Jaú, Jaú, São Paulo
  - São José do Rio Preto, São José do Rio Preto, São Paulo